CLINICAL TRIAL: NCT04592367
Title: Rekonstruktion af Forreste korsbånd Hos +30-årige Vurderet Ved Patient Reported Outcome Measures(PRO)
Brief Title: Reconstruction of the Anterior Cruciate Ligament(ACL-R) in the 30+-Year Old Assessed by Patient Reported Outcome Measures(PRO) Using the Nationwide Danish Knee Ligament Reconstruction Registry
Status: Completed | Type: Observational
Sponsor: Region Zealand (Other)
Responsible Party: Principal Investigator, Jesper Glerup, Research Student, Region Zealand
Other Study IDs: PRO-4ACL
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Cruciate Ligament Rupture
Keywords: ACL,; PRO; PROM; age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Patient age at time of procedure of reconstruction of ACL — Primary reconstruction of ACL with no other concomitant ligament reconstructions. Treatment of cartilage og meniscal injury may be a part of the procedure

SUMMARY:
The purpose of the study is to evaluate the efficacy of primary ACL-R in patients 30 years of age or older using PRO. The PRO used are Knee Osteoarthritis Outcome Score(KOOS) and Tegner score. The Danish Knee Ligament Reconstruction Registry has data including more than 31,000 primary ACL-R performed in the period from 2005 to 2018, of which approximately a little less than 40% are performed in patients 30 years or older.

Traditionally, ACL-R has been used for the active, younger patients with the purpose of returning to their pre-injury level of activity. The increasing activity level and the desire to stay active among some patients in their fourth decade, and later, possibly increases the demands of the reconstructed ACL in this group. The aim is to investigate the PRO in this group of patients and compare them with the PRO of patients younger than 30 years of age. The study may help orthopedic surgeons counselling patients 30 years of age or older when deciding to perform an ACL-R.

The study's hypothesis is, that the overall benefit from ACL-R is equal but the patients 30 years of age or older has a worse baseline and as an implication of that worse PRO one year after the ACL-R.

DETAILED DESCRIPTION:
Quality Assurance Plan: Clinical data reported by orthopedic surgeons at public and private hospitals, while patients undergoing ACL-R report PRO.

Source Data Verification with the Danish National Central Person Registry. Degree of completeness compared to Central Person Registry is approximately 85%.

Data dictionary provided by the data manager at RKKP - "Regionernes Kliniske Kvalitetudviklingsprogram" - Regional Clinical Quality Development Program. Patients are recruited when the ACL-R is performed, and approximately 35% report PRO 1 year after surgery. Data collection, data management and the extract from the Danish Knee Ligament Reconstruction Registry is performed by the Regional Clinical Quality Development Program. Data analysis done with support from statistician from "Region Sjælland" - Region Zealand. Sample Size Assessment not done. The cohort size is the largest we can get from the registry. The estimated number of patients 30 years of age or older with complete PROs is 2,600 men and 1,600 women. This estimation is based on the numbers from the annual report of 2019 from the Danish Knee Ligament Reconstruction Register, which states that 7,368 men and 4,656 women 30 years of age or older has undergone the procedure from 2005-2018. We expect that they report PROs as frequently as the entire cohort, which is approximately 35%. Patients with missing data will be described in table 3 and not used in table 2.

The study will present five tables.

Flowchart: Cohort size, excluded patients, patients with missing values, patients in each age group

Table 1: Descriptive statistics of the cohort with reported PRO stratified in three strata (0-14 years of age, 15-29 years of age or 30 years of age or older) with information about gender, age, previous surgery in the knee, activity at time of injury, operational technique and cartilage and meniscal status.

Table 2: Unpaired t-test if data shows normal distribution, otherwise Mann-Whitney, by change in KOOS from before surgery to one year after surgery, overall KOOS one year after surgery, Tegner one year after surgery, and Tegner from preoperatively to one year after surgery

Table 3: Descriptive statistics of population lost during follow-up

Table 4: Multivariate analysis for primary outcome

Sampling Method: Consecutive patients. Patients are enrolled into the registry when the ACL-R is performed. The completeness of registry depends on physicians' reporting of pre-, intra- and postoperative findings and patients' reporting of PROs.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving primary reconstruction of the ACL in the period 1st of January 2005 to 31st of December 2018

Exclusion Criteria:

* Multi Ligament Surgery
* Revision surgery of ACL

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is the entire Danish population. The completeness of registry, the epidemiology of ACL-rupture and ACL-R decides the composition of the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 30487 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in KOOS | From before surgery, but after injury, to one year after surgery

SECONDARY OUTCOMES:
Total KOOS | One year after surgery
Total Tegner score | One year after surgery
Change in Tegner score | From before surgery, but after injury, to one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Glerup, Medical Student, Principal Investigator — Region Zealand; Jakob Klit, MD, PhD, Associate Professor, Principal Investigator — Region Zealand
Locations (1):
- Department of Orthopedic Surgery, Køge, Region Zeland, Denmark

IPD SHARING:
Plan to Share IPD: No